CLINICAL TRIAL: NCT06158464
Title: The Effectiveness of a Functional Capacity Evaluation (FCE) on the Return-to-work Process in Belgium: a Randomized Controlled Trial
Brief Title: The Effectiveness of a Functional Capacity Evaluation Among Persons on Sick Leave or Work Disability
Acronym: FCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Haute École Léonard de Vinci (Unknown); National Institute for Health and Disability Insurance (NIHDI), Belgium (Unknown)
Responsible Party: Principal Investigator, Lode Godderis, prof. dr. (MD), KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCE-study
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Sick Leave; Absenteeism; Return to Work
Keywords: return-to-work; functional capacity evaluation; randomized controlled trial; workability; occupational therapy

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial will be set up (RCT). For this purpose, 10 consulting physicians, 30 occupational therapists, and 200 persons on incapacity will be recruited. Then, persons on sick leave/work disability are randomly divided into two groups: 1) Persons in the control group receive care-as-usual without modifications. 2) Persons in the intervention group receive usual care and a functional capacity evaluation (FCE). Both groups are asked to complete questionnaires at baseline, and after 3,6, and 9 months. Primary outcome is the difference in workability at 6 months follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care-as-usual (No Intervention): In standard care, persons on sick leave/work disability are invited by the medical advisor for a consultation. If the patient is allocated to the control group (or if the patient did not agree to participate in the study), the medical advisor takes decisions based on the information at his disposal, e.g. start a return-to-work trajectory, to temporarily prolong sickness absence and disability, or to confirm definitive work disability. If they agree to participate, they are asked to complete four questionnaires: at baseline, at 3 months, 6 months, and 9 months.
- Care-as-usual supplemented by a Functional Capacity Evaluation (Experimental): In the intervention group, participants are referred to an occupational therapist to receive an FCE. Afterwards, the occupational therapist completes a standardized FCE-template, and conveys these recommendations to the medical advisor. This template includes a list of ICF categories important to the work context. The conclusion of the FCE includes: 1) The facilitators and barriers related to work-related physical, cognitive or psychological functioning, or related to environmental and/or psychosocial factors. 2) A recommendation on the current or last occupation or a reference occupation with or without adaptation and/or on reorientation, training, coaching.
  Based on the FCE results, the medical advisor can adapt his advice and communicate to the person on sick leave/work disability to advise him/her, or refer the person on sick leave/work disability to other partners (such as VDAB, FOREM, Actiris, or the RTW-coordinator).
  Interventions: Other: Functional Capacity Evaluation

INTERVENTIONS:
Other: Functional Capacity Evaluation — In a FCE, an occupational therapist will evaluate a patient's ability to perform work-related tasks, using a battery of tests. Depending on the circumstances, he/she will for instance test fatigue, ask the patient to kneel, lift objects, or assess concentration. This assessment lasts ± 4 hours and includes physical tests and tests related to the (previous or reference) profession of the client. This means that an explicit match is made between the functional capacities of the patient (what is he/she capable of) and the demands of a certain job (what is he/she expected to do). Following this assessment, the occupational therapist will explain the results of this assessment to the patient. The evaluation will therefore take place during one or two visits.
  Arms: Care-as-usual supplemented by a Functional Capacity Evaluation

SUMMARY:
The goal of this clinical trial is to evaluate Functional Capacity Evaluations in persons on sick leave or work disability. The main questions it aims to answer are:

* What is the impact of FCE on the person on sick leave/work disability (quantitative)
* What is the impact of FCE on the decision-making process by the medical advisor? (qualitative)
* What is the usability, feasibility and quality of FCE for the medical advisor, occupational therapist, mediators of the regional services, and return-to-work coordinators? (qualitative)

This is a randomized controlled trial (RCT). Participants in the control group will receive care-as-usual by the medical advisor. Participants in the intervention group will receive an FCE on top of care-as-usual. This is performed by an occupational therapist in their region, and a report of the FCE is delivered to the medical advisor. Both groups are asked to complete questionnaires at baseline, and after 3,6, and 9 months.

Researchers will compare questionnaire results from participants in the control and intervention group, to see if their workability (primary outcome), steps to return to work, expectations to return to work, return to work beliefs, time until (partial) reintegration, self-efficacy in return to work, pain scale, and illness perception (secondary outcomes) are affected differently.

DETAILED DESCRIPTION:
This research project on the use of Functional Capacity Evaluations (FCE) within the context of benefit insurance in Belgium falls under the joint control of the National Institute for Sickness and Disability Insurance (RIZIV), the Haute École de Leonard Vinci and KU Leuven . KU Leuven hereby acts as the study's principal, but together with RIZIV and Haute École determines the objectives of the study as joint controllers.

An FCE consists of the evaluation of functional capacities based on medical reporting, observations and/or a series of standardised tests performed by an occupational therapist. This evaluation can give socially insured persons and medical advisors of the mutualities more insight into the participation possibilities of the socially insured person in function of the previous or next job. To date, the advisory doctor does not yet have the opportunity to have these evaluations carried out in Belgium. The aim of this study is therefore to examine the impact of these FCEs with regard to people on incapacity for work who meet the following conditions:

1. Belgian citizens on sick leave or work disability who meet the criteria determined by the article 100§1 and 100 §2 of the coordinated law of 14 July 1994, or by article 19 and/or 20 of the RD 20 July 1971.
2. The person's medical situation is stabilised (no significant evolution due to illness, procedure, treatment)
3. It is not a purely mental/psychiatric disorder
4. From the point of view of the consulting physician, there is a lack of consistent information on the capacity to return to work
5. Inclusion takes place from the 6th month of incapacity
6. The person is of working age: 18-65 years

In this RCT, 10 consulting physicians, 30 occupational therapists, and 200 persons on incapacity will be recruited. Then, persons on sick leave/work disability are randomly divided into two groups: 1) Persons in the control group receive the usual counselling by the medical advisor. 2) Persons in the intervention group receive usual care and an FCE. In the latter group, the person on sick leave is matched by the researchers to an occupational therapist in his region, and is invited to a FCE. After the evaluation, the person reviews the results with the occupational therapist, and a report of the FCE is provided to the medical advisor. Finally, the person is contacted by the medical advisor if they wish to take certain actions as a result of the FCE report. To measure the impact of the FCE, the intervention and control groups thereby complete a questionnaire at four points in time: at baseline, after 3 months, after 6 months, and after 9 months. This questionnaire is composed of validated instruments, and in addition to background characteristics, it questions work ability, self-efficacy, expectations of returning to work, any (steps taken to) return to work, pain intensity, illness perception, and beliefs regarding returning to work.

As a second objective, the impact on the medical advisors' (and other parties') decision-making process will be investigated through qualitative interviews and focus groups. To this end, a process evaluation will be conducted. This includes an examination of the implementation of the study, the usability, feasibility and quality of FCEs and their reporting, and the underlying causal mechanisms of the intervention. Using interviews and focus groups with medical advisors the impact of the FCE on the decision-making process will be investigated. Using interviews with occupational therapists, return-to-work coordinators and mediators of the regional services the usability, feasibility and quality of the FCE will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* persons on sick leave or work disability (according to Belgian law)
* The person on sick leave/work disability is affected by an illness/injury that is considered stabilized (no significant medical evolution of the disease, nor a medical procedure or acute treatment is expected).
* The illness/injury of the person on sick leave/work disability is not mainly a mental/psychiatric disorder.
* From the point of view of the medical advisor, there is a lack of consistent information on the person on sick leave/work disability's capacity to return-to-work.
* Inclusion takes place from the 6th month of incapacity for work.
* The person on sick leave/work disability is of working age (18-65).

Exclusion Criteria:

* In the case of an accident at workplace, the medical condition of the person on sick leave/work disability has not yet been declared consolidated, meaning that the condition does not progress significantly, either naturally or with treatment.
* The medical advisor of the mutual health insurance is expecting in the near future: 1) a spontaneous return to work (total or partial), 2) a registration as a job-seeker, or 3) an end of the recognition of the work disability.
* The person on sick leave/work disability is pregnant.
* The medical advisor of the mutual health insurance perceives the person on sick leave/work disability does not have sufficient work capacity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Workability | measured at baseline, and 3, 6 and 9 months post baseline
  The single-item first WAI (Work Ability Index) question is a self-report question in which the person rates his "current work ability compared with the lifetime best", with a score of 0 ("completely unable to work") up to 10 ("work ability at its lifetime best").

SECONDARY OUTCOMES:
Self-efficacy in the context of return-to-work | measured at baseline, and 3, 6 and 9 months post baseline
  The self-efficacy return to work scale is a 10 item self-report questionnaire consisting of three subdomains of self-efficacy: (1) ability to cope with pain, (2) ability to obtain help from supervisor, and (3) ability to obtain help from co-workers. (Brouwer et al., 2009, 2010). There are five response options; for each item the person is asked to rate his/her confidence on a five-point scale (0 = not at all certain, 4 = completely certain). Subscores and an overall score (i.e., summative score) can be obtained, with higher scores indicating better return-to-work self-efficacy.
Expectations to return-to-work | measured at baseline, and 3, 6 and 9 months post baseline
  A single-item question "To what extent do you think you will return to work?" with the 4 response options: 1 (to a low degree); 2 (to a certain degree); 3 (to a high degree); 4 (do not know)
Steps to return-to-work | measured at baseline, and 3, 6 and 9 months post baseline
  The participants indicate which steps they have undertaken in their return-to-work, multiple answers are possible. Answers range from following training programmes, looking for jobs, undergoing work-oriented rehabilitation, to returning to work at a new or former employee.
Pain scale | measured at baseline, and 3, 6 and 9 months post baseline
  The Graded Chronic Pain Scale Revised (GCPS-R) is a 5-item self-report questionnaire assessing (1) current pain, (2) limitations in life or work abilities, (3) general pain, (4) enjoyment of life, (5) interference with general activity. For items 1 and 2, responses options are Never/Some days/Most days/Everyday, for items 3 responses options are the following: from 0 (No pain) to 10 (Pain as bad as you can imagine) while for items 4 and 5 responses options are the following : from 0 (does not interfere) to 10 (completely interferes).
Illness perception | measured at baseline, and 3, 6 and 9 months post baseline
  The Brief IPQ has nine items, it is designed to measure patients' cognitive and emotional representations of their illness including consequences (item 1), timeline (item 2), personal control (item 3), treatment control (item 4), identity (item 5), coherence (item 6), concern (item 7), emotional response (item 8), and causes (item 9) (Broadbent et al., 2006). All of the items except the causal question are rated using a 0-to 10 response scale. Increases in item scores represent linear increases in the dimension measured.
Return-to-work beliefs | measured at baseline, and 3, 6 and 9 months post baseline
  The RTW Beliefs questionnaire is composed of 12 items divided into four subscale of general direct measures: intention (i.e., "I expect to/want to/intend to …"), attitude (i.e., "RTW is for me: harmful-beneficial/ good-bad/pleasant-unpleasant/worthless-useful"), subjective norms (i.e., "It is expected of me that I should … /I feel under social pressure to … /People who are important to me want me to …" ) , and perceived behavioural control (i.e., "I'm confident that I could … / for me RTW is (easy-difficult).

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (8):
  - MC Hainaut, Anderlues
  - LM Plus Antwerpen, Antwerp
  - Helan/Medisch kabinet Genk, Genk
  - CM Gent, Ghent
  - CM Vlaams-Brabant, Leuven
  - MC Liège, Liège
  - CM Oostende, Ostend
  - Mutsoc Luxembourg, Saint-Hubert

IPD SHARING:
Plan to Share IPD: Yes
Apart from the researchers, the National Institute for Health and Disability Insurance (NIHDI) will have access to the pseudonymised questionnaire data, as specified in a GDPR-contract. Selected questionnaire data as well as the FCE-results will be available to the occupational therapists, the medical advisor, the return-to-work coordinator, and the mediator of the regional services.
Supporting Information: Study Protocol, CSR
Time Frame: starting december 2024
Access Criteria: pseudonymized raw data